CLINICAL TRIAL: NCT05496465
Title: A Single-Dose, Randomized, Placebo-Controlled, Cross-Over Study of the Safety and Efficacy of Intranasal Epinephrine After Administration of ARS -1 in Subjects With Frequent Urticaria Flares
Brief Title: Safety and Efficacy of Intranasal Epinephrine After Administration of ARS -1 in Subjects With Frequent Urticaria Flares
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARS Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RELIEF-CSU1
Record Dates: First submitted 2022-04-27; First posted 2022-08-11 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Urticaria
MeSH Terms: conditions — Urticaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ARS-1 1mg (Active Comparator): 1 mg per 100 µL dose of ARS-1
  Interventions: Drug: ARS-1
- ARS-1 2mg (Active Comparator): 2 mg per 100 µL dose of ARS-1
  Interventions: Drug: ARS-1
- Placebo (Placebo Comparator): Placebo (100 µL)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARS-1 — A single treatment of ARS-1.
  Arms: ARS-1 1mg; ARS-1 2mg
Drug: Placebo — A single treatment of placebo nasal spray
  Arms: Placebo

SUMMARY:
Determine the effect of ARS-1 on a patient reported pruritus/hive score

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female subject between the ages of 18 and 65 years.
* 2. Clinically diagnosed urticaria with acute symptom flares at least two (2) times a week while on a chronic treatment.
* 3. Body weight more than 30 kg and body mass index between 18 and 34 kg/m².
* 4. Has no medical history of hypertension and cardiovascular disease in the last 10 years.
* 5. At screening, has stable vital signs.
* 6. If female, is not pregnant or breastfeeding.
* 7. If male (with or without vasectomy), agree to the use of highly effective contraceptive methods at screening until 7 days after the last day of study drug.

  8. Is able to communicate clearly with the Investigator and staff. 9. Provide written informed consent prior to participating in the study.

Exclusion Criteria:

* 1. History of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease.
* 2. Patients receiving beta blocker due to potential interaction with the study drug.
* 3. Prior nasal fractures, severe nasal injuries or history of nasal disorders.
* 4. Clinically significant medical condition or physical exam finding.
* 5. Abnormal cardiovascular exam at screening including any prior history of myocardial infarction or clinically significant abnormal ECG.
* 6. Mucosal inflammatory disorders.
* 7. Significant traumatic injury or major surgery within 30 days prior to study screening.
* 8. Has donated blood or had an acute loss of blood (>50 mL) during the 30 days before study drug administration.
* 9. Known hypersensitivity to any compound in the test product.
* 10. Participated in a clinical trial within 30 days prior to the first dose of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Effect of ARS-1 versus placebo based on a patient reported pruritus/hive score | Assessment will start from 1 hour pre-dose to 120 (± 10 min) minutes after dosing.
  Assess time to effect and duration of effect on acute flares associated with urticaria based on a patient reported pruritus/hive score.

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Tanimoto, MD, PhD, Study Director — ARS Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio